CLINICAL TRIAL: NCT05675332
Title: Effects of Stereotype Threat on Impulsivity and Its Relation to Alcohol Use in African Americans: An fMRI Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Uraina S Clark, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 19-0250; R01AA028023 (NIH)
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no stress exposure (Placebo Comparator): no threat stress
  Interventions: Behavioral: Task-based behavioral intervention
- stress exposure (Active Comparator): exposure to stress threat
  Interventions: Behavioral: Task-based behavioral intervention

INTERVENTIONS:
Behavioral: Task-based behavioral intervention — Brief behavioral intervention is absent of stressors.
  Arms: no stress exposure
Behavioral: Task-based behavioral intervention — Brief behavioral intervention involves interacting with common everyday types of stress.
  Arms: stress exposure

SUMMARY:
The purpose of this study is to investigate the behavioral and neural correlates of stress exposure. Results from this study will enrich the understanding of how sociocultural, behavioral, and neural factors combine to influence alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 35 years of age (inclusive);
* Fluent in English;
* Right-handed

Exclusion Criteria:

* Younger than 21 years of age;
* Left-handed

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen-level dependent (BOLD) signal | Baseline
  Blood oxygen-level dependent (BOLD) signal in brain regions of interest (ROI) measured using fMRI
Resting-state functional connectivity in brain regions | Baseline
  Resting-state functional connectivity - brain activity measured using fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Uraina Clark, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD